CLINICAL TRIAL: NCT00005327
Title: Prevention of Cerebral Infarction in Sickle Cell Anemia - Comprehensive Sickle Cell Center
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4117; P60HL048484 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2017-03

CONDITIONS: Anemia, Sickle Cell; Blood Disease; Cerebrovascular Disorders; Cerebrovascular Accident
MeSH Terms: conditions — Anemia, Sickle Cell; Hematologic Diseases; Cerebrovascular Disorders; Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To conduct a prospective study aimed at the early detection and treatment of cerebral vascular disease prior to irreversible brain injury in young children with sickle cell anemia (SCA).

DETAILED DESCRIPTION:
BACKGROUND:

Cerebral infarction is a major contributor to childhood morbidity and mortality in sickle cell anemia (SCA)

DESIGN NARRATIVE:

The investigators tested the hypotheses that young children with SCA experienced a variable period of asymptomatic progressive central nervous system (CNS) vasculopathy prior to cerebral infarction; that pre-infarct CNS vasculopathy could be identified by non-invasive imaging techniques:MRI, magnetic resonance angiography (MRA), and transcranial Doppler (TCD); and that therapeutic intervention at this stage of the disease could significantly reduce the subsequent occurrence of cerebral infarction. MRI, MRA, TCD, and standardized neurologic and psychometric examinations were performed yearly in a cohort of homozygous Hb SS children enrolled at 2-4 years of age. Subjects without MRI evidence of cerebral infarction who had significant cerebral vasculopathy (cerebral arterial stenosis on MRA and/or elevated blood flow velocity on TCD) were randomized to receive either no therapy or chronic transfusion therapy, in order to determine the risk of subsequent cerebral infarction in untreated subjects with these abnormalities, and the extent to which transfusion therapy could significantly reduce the risk. Subjects with evidence of prior cerebral infarction on MRI, whether symptomatic or asymptomatic, were randomized to receive either chronic transfusion therapy alone ('standard therapy') or chronic transfusion therapy plus ticlopidine, in order to determine whether ticlopidine could significantly increase the efficacy of standard therapy in preventing recurrent cerebral infarction in SCA. Subjects with prior cerebral infarction were also offered the option of bone marrow transplantation if an HLA-identical non-SS sibling donor was available.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-04 (Actual); Primary Completion 1998-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darleen Powars — University of Southern California

REFERENCES:
- [Background] Powars DR, Conti PS, Wong WY, Groncy P, Hyman C, Smith E, Ewing N, Keenan RN, Zee CS, Harold Y, Hiti AL, Teng EL, Chan LS. Cerebral vasculopathy in sickle cell anemia: diagnostic contribution of positron emission tomography. Blood. 1999 Jan 1;93(1):71-9. PMID 9864148
- [Background] Powars DR. Management of cerebral vasculopathy in children with sickle cell anaemia. Br J Haematol. 2000 Mar;108(4):666-78. doi: 10.1046/j.1365-2141.2000.01912.x. No abstract available. PMID 10792268